CLINICAL TRIAL: NCT00401050
Title: A Randomized Clinical Trial Comparing Two Chiropractic Protocols for Patellofemoral Pain Syndrome: a Pilot Study
Brief Title: Comparison Study of Two Chiropractic Treatment Protocols for Knee Pain Due to Patellofemoral Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cleveland Chiropractic College (Other)
Responsible Party: James W. Brantingham, DC, PhD, Cleveland Chiropractic College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 06-15-06
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2010-04-20 (Estimated); Status verified 2010-04

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: patellofemoral pain syndrome; chiropractic; knee pain; chiropractic manipulation; Graston Instrument Soft Tissue Mobilization(GISTM)
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: chiropractic manipulative therapy
Procedure: knee exercises
Procedure: Graston Instrument Soft Tissue Mobilization (GISTM)

SUMMARY:
The purpose of this study is to compare outcomes of combined chiropractic care in anterior knee pain patients with patellofemoral pain syndrome.

DETAILED DESCRIPTION:
Exercise is standard of care for PFPS but gives limited pain reduction and functional improvement. Previous manipulative therapy for PFPS (with and without exercise) has been limited to the patellofemoral joint alone. However, literature suggests additional manipulative therapy with exercise and soft-tissue treatment may give a better outcome. Further research is needed.

Therefore, this project is a pilot study to inform a future randomized controlled trial to determine if chiropractic adjusting of the full lower extremity (lumbosacral through foot) combined with exercise and soft tissue treatment (Protocol and group A) is superior to chiropractic adjusting of the knee (alone) combined with exercise and soft tissue treatment (Protocol and group B) in the treatment of patellofemoral pain syndrome. We will use the Anterior Knee Pain Scale (AKPS) and Visual Analogue Scale (VAS) as valid and reliable primary outcome measures, a functional measure (step-ups, step-downs and squats) and a Patient Satisfaction Scale (PSS - discharge or refer) as secondary outcome measures. This study will help establish the feasibility of conducting quality research at Cleveland Chiropractic College Los Angeles.

In this pilot study there will be two groups of 10 subjects each

1. Group A will receive CMT to the knee only, exercise and soft tissue treatment (Graston Instrument Soft Tissue Mobilization hereafter GISTM)
2. Group B will receive CMT to the lumbosacral, sacroiliac and (all) lower extremity joints, exercise and soft tissue treatment (GISTM).

Enrolled subjects will receive a total of 6 treatments. The primary endpoint will be a 2 month follow-up after the 6th treatment.

ELIGIBILITY:
Inclusion Criteria:

* anterior, peri or retropatellar knee pain >3 months from at least two of the following: prolonged sitting, stair-climbing, squatting, running, kneeling, and hopping/jumping or overuse activities. Pain is relieved by rest.
* insidious onset of symptoms unrelated to a traumatic incident; and
* presence of pain on palpation of the patellar facets, on step down from a 25-cm step, or during a double-legged squat
* other disorders such as OA, instability or medial meniscus injury must be ruled out
* X-ray or MRI findings not required. There is no clear correlation between severity of complaints and arthroscopic or radiologic findings
* A VAS-Worst pain of ≥ 5.0; a AKPS of ≥ 50.This reflects the current probability that less PFPS patients with less severity currently consult chiropractors for this disorder

Exclusion Criteria:

* Patellar subluxation/dislocation
* meniscal injuries
* intra-articular pathology (ACL injury, etc)
* ligament laxity
* Osgood-Schlatters
* Sinding-Larsen-Johanson syndrome
* knee joint effusion
* previous surgery on patellofemoral joint
* illiteracy/inability to understand and answer questionnaires
* inability to attend all treatment sessions
* true locking of knee joint
* a neurological disorder that influences gait
* if taking medication, amount will be diarized - otherwise not allowed
* foot orthotics allowed if already worn
* arthritidies
* bursitis
* patellar tendonitis
* older subjects > 45 years of age
* subjects < 18 years of age
* those that begin marked ↑ in physical activity during the course of the trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2006-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Anterior Knee Pain Scale (AKPS)before treatment, after last treatment and at 2 month follow up | Baseline, 6th Treatment, 2 Month Follow-Up
Visual Analogue Scale (VAS) before treatment, after last treatment and at 2 month follow up | Baseline, 6th Treatment, 2 Month Follow-Up

SECONDARY OUTCOMES:
a functional measure (step-ups, step-downs and squats) before treatment, after last treatment and at 2 month follow up | Baseline, 6th Treatment, 2 Month Follow-Up
Patient Satisfaction Scale at 2 month follow up only | Baseline, 6th Treatment, 2 Month Follow-Up

CONTACTS AND LOCATIONS:
Overall Officials: James W. Brantingham, D.C., PhD., Principal Investigator — Cleveland Chiropractic College Los Angeles
Locations (1):
- Cleveland Chirpractic College Los Angeles, Los Angeles, California, United States